CLINICAL TRIAL: NCT00160199
Title: Evaluation of Safety and Efficacy of PROMETRIUM® Capsules in Induction of Secretory Conversion of Endometrium and Withdrawal Bleeding in Subjects With Secondary Amenorrhea
Brief Title: Safety and Efficacy of PROMETRIUM® Capsules in Induction of Secretory Conversion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Cindy Lane, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S168.4.002
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2010-06-02 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-06

CONDITIONS: Secondary Amenorrhea
Keywords: To collect additional data on 300 and 400 mg doses of PROMETRIUM in women with secondary amenorrhea
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: PROMETRIUM® 300 mg
- 2 (Active Comparator)
  Interventions: Drug: PROMETRIUM® 400 mg

INTERVENTIONS:
Drug: PROMETRIUM® 300 mg — 300 mg (3x100mg capsules) by mouth once daily at bedtime for 10 days X 3 cycles
  Arms: 1
Drug: PROMETRIUM® 400 mg — 400 mg (4x100mg capsules) by mouth once daily at bedtime for 10 days X 3 cycles
  Arms: 2

SUMMARY:
To evaluate the efficacy and safety of 300 mg and 400 mg doses of PROMETRIUM® capsules in women of reproductive age with secondary amenorrhea

ELIGIBILITY:
Inclusion Criteria:

* Women with secondary amenorrhea
* Normal serum Dehydroepiandrosterone (DHEA), prolactin, testosterone, Thyroid Stimulating Hormone (TSH) and thyroxine

Exclusion Criteria:

* Primary amenorrhea
* Other medical conditions resulting in amenorrhea (e.g. Asherman's syndrome)
* Peanut allergy
* Allergy to progestational steroids

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2004-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (42):
- United States (42):
  - Site 29, Mobile, Alabama
  - Site 41, Montgomery, Alabama
  - Site 26, Tucson, Arizona
  - Site 5, Jonesboro, Arkansas
  - Site 39, Carmichael, California
  - Site 17, Encinitas, California
  - Site 10, San Diego, California
  - Site 42, Avon, Connecticut
  - Site 3, Groton, Connecticut
  - Site 22, New Britian, Connecticut
  - Site 9, Waterbury, Connecticut
  - Site 37, West Hartford, Connecticut
  - Site 14, Aventura, Florida
  - Site 40, Clearwater, Florida
  - Site 1, West Palm Beach, Florida
  - Site 30, West Palm Beach, Florida
  - Site 46, Atlanta, Georgia
  - Site 43, Powder Springs, Georgia
  - Site 36, Champaign, Illinois
  - Site 12, Chicago, Illinois
  - Site 6, Baton Rouge, Louisiana
  - Site 7, Baltimore, Maryland
  - Site 2, St Louis, Missouri
  - Site 16, Reno, Nevada
  - Site 45, New York, New York
  - Site 23, New Bern, North Carolina
  - Site 15, Winston-Salem, North Carolina
  - Site 28, Winston-Salem, North Carolina
  - Site 33, Cincinnati, Ohio
  - Site 32, Erie, Pennsylvania
  - Site 47, Hershey, Pennsylvania
  - Site 44, Philadelphia, Pennsylvania
  - Site 38, Pottstown, Pennsylvania
  - Site 13, Greenville, South Carolina
  - Site 8, Conroe, Texas
  - Site 11, Corpus Christi, Texas
  - Site 27, Houston, Texas
  - Site 34, Houston, Texas
  - Site 24, San Antonio, Texas
  - Site 35, Salt Lake City, Utah
  - Site 19, Norfolk, Virginia
  - Site 4, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in 42 centers in US between November 2004 and February 2009. Before the randomization, subjects were evaluated for eligibility. In total 240 subjects were randomized.
Pre-assignment Details: The Baseline characteristics are presented using the Full Analysis Sample (FAS) to be online with the Efficacy analysis results.
Period: Overall Study
Arm/Group | Prometrium 300 mg/Day | Prometrium 400 mg/Day
Started | 122 | 118
Completed | 98 | 81
Not Completed | 24 | 37
Not completed — Adverse Event | 5 | 14
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 7 | 7
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Administrative | 0 | 1
Not completed — Protocol Violation | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prometrium 300 mg/Day | Prometrium 400 mg/Day | Total
Number analyzed (Participants) | 107 | 99 | 206
Age Continuous [Mean (Standard Deviation); unit: years] — The participant flow chart was done on all Randomized subjects set (i.e. subjects who received at least one dose of open-label study medication) . The baseline results are presented on the Full Analysis set (i.e. subjects randomized with at least one post-baseline evaluable efficacy assessment).
  years | 29.2 (6.63) | 28.7 (6.35) | 29.0 (6.49)
Sex: Female, Male [Count of Participants; unit: Participants] — The participant flow chart was done on all Randomized subjects set (i.e. subjects who received at least one dose of open-label study medication) . The baseline results are presented on the Full Analysis set (i.e. subjects randomized with at least one post-baseline evaluable efficacy assessment).
  Participants
    Female | 107 | 99 | 206
    Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — The participant flow chart was done on all Randomized subjects set (i.e. subjects who received at least one dose of open-label study medication) . The baseline results are presented on the Full Analysis set (i.e. subjects randomized with at least one post-baseline evaluable efficacy assessment).
  participants
    United States | 107 | 99 | 206

OUTCOME MEASURES:

1. Primary Outcome: Secretory Conversion of the Endometrium
Description: Endometrial biopsy results were classified as : Secretory (Complete or partial), Non-secretory, Unable to determine or Unknown after an evaluation of morphologic criteria.
Time Frame: End of the study (Days 85)
Population: The analysis was done on the Full Analysis Sample defined as subjects who received at least one dose of treatment and with at least one post-baseline evaluable efficacy assessment. Only summary statistics were generated.
Measure: Number; unit: participants
Arm/Group | Prometrium 300 mg/Day | Prometrium 400 mg/Day
Number analyzed (Participants) | 107 | 99
participants
  Secretory | 23 | 28
  Non-Secretory | 70 | 53
  Unable to determine | 7 | 9
  Unknown | 4 | 2

2. Primary Outcome: Number of Subjects With Withdrawal Bleeding
Description: This measure is the number of subjects with withdrawal bleeding using Last Observation Carried Forward (LOCF) after first and second cycle.
Time Frame: After first and second cycle (cycle=28 days)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Prometrium 300 mg/Day | Prometrium 400 mg/Day
Number analyzed (Participants) | 107 | 99
participants | 93 | 90

3. Secondary Outcome: Maximum Intensity of Withdrawal Bleeding After Any Cycle
Description: The intensity of withdrawal bleeding was classified by: None, Spotting, Light, Moderate, Heavy
Time Frame: Duration of withdrawal bleed
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Prometrium 300 mg/Day | Prometrium 400 mg/Day
Number analyzed (Participants) | 107 | 99
participants
  None | 13 | 8
  Spotting (Intermittent Staining) | 10 | 3
  Light (Slight amount-continuous staining) | 18 | 14
  Moderate (Modest amount-continuous staining) | 25 | 40
  Heavy (Large amount-heavy clots) | 40 | 33

4. Secondary Outcome: The Duration of Withdrawal Bleeding After the First Treatment Cycle
Description: The numbers of days the subjects actually bled after the end of the first treatment cycle.
Time Frame: End of the first cycle of treatment (cycle=28 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Prometrium 300 mg/Day | Prometrium 400 mg/Day
Number analyzed (Participants) | 107 | 99
Days | 4.0 (2.03) | 3.8 (1.88)

5. Secondary Outcome: The Duration of Withdrawal Bleeding After Second Treatment Cycle
Description: The numbers of days the subjects actually bled after the end of the second treatment cycle
Time Frame: End of the second cycle of treatment (cycle=28 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Prometrium 300 mg/Day | Prometrium 400 mg/Day
Number analyzed (Participants) | 107 | 99
Days | 3.5 (2.15) | 3.8 (1.62)

6. Secondary Outcome: Time to Withdrawal Bleeding After First Treatment Cycle
Description: The number of days between the first cycle of treatment and the withdrawal bleeding.
Time Frame: End of the first cycle of treatment (cycle=28 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Prometrium 300 mg/Day | Prometrium 400 mg/Day
Number analyzed (Participants) | 107 | 99
Days | 1.9 (1.89) | 2.2 (1.81)

7. Secondary Outcome: Time to Withdrawal Bleeding After Second Treatment Cycle
Description: The number of days between the second cycle of treatment and the withdrawal bleeding
Time Frame: End of the second cycle of treatment (cycle=28 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Prometrium 300 mg/Day | Prometrium 400 mg/Day
Number analyzed (Participants) | 107 | 99
Days | 1.6 (1.99) | 2.21 (1.72)

ADVERSE EVENTS:
Time Frame: The adverse events presented were collected from start of drug treatment to the end of the treatment period.
Description: The safety analysis is presented on the safety sample meaning the number of patients who were randomized and received at least one dose of study medication.
Arm/Group | Prometrium 300 mg/Day | Prometrium 400 mg/Day
Serious Adverse Events (participants affected / at risk) | 2/113 | 1/107
Other Adverse Events (participants affected / at risk) | 72/113 | 70/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prometrium 300 mg/Day (N=113) | Prometrium 400 mg/Day (N=107)
Adnexa uteri mass (Reproductive system and breast disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prometrium 300 mg/Day (N=113) | Prometrium 400 mg/Day (N=107)
Acnes (Skin and subcutaneous tissue disorders) | 8 | 7
Asthenic conditions (General disorders) | 11 | 7
Breast signs and symptoms (Reproductive system and breast disorders) | 8 | 5
Flatulence Bloating and distension (Gastrointestinal disorders) | 6 | 5
Fungal infection NEC (Infections and infestations) | 9 | 6
Gastrointestinal and Abdominal Pains (excl oral and throat) (Gastrointestinal disorders) | 9 | 6
Headaches NEC (Nervous system disorders) | 13 | 9
Musculoskeletal and connective tissue signs and symptoms NEC (Musculoskeletal and connective tissue disorders) | 6 | 5
Nausea and Vomiting (Gastrointestinal disorders) | 15 | 9
Neurological signs and symptoms NEC (Nervous system disorders) | 6 | 8
Upper respiratory tract infections (Infections and infestations) | 13 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Independent analysis and/or publication of these data by the investigator or any member of his/her staff are not permitted without prior written consent of Solvay Pharmaceuticals,Inc. Written permission will be contingent on the review by Solvay Pharmaceuticals, Inc. of the statistical analysis and manuscript and providing for non-disclosure of Solvay Pharmaceuticals, Inc. confidential or proprietary information.